CLINICAL TRIAL: NCT01054482
Title: A Randomized Phase II Study Preoperative Chemotherapy Versus Preoperative Concurrent Chemoradiotherapy for Patients With Locally Advanced Non-Small Cell Lung Cancer
Brief Title: Pre-operative Chemotherapy Versus Concurrent Chemoradiotherapy in Locally Advanced Non-small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: The First Affiliated Hospital of Guangzhou Medical College, Guangzhou Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FAHG20070218
Record Dates: First submitted 2010-01-21; First posted 2010-01-22 (Estimated); Last update posted 2010-02-02 (Estimated); Status verified 2007-01

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Neoadjuvant chemotherapy; neoadjuvant chemoradiotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pre-operative chemotherapy (Experimental): Docetaxel 75 mg/m2 + Carboplatin AUC(area under the curve)=6 on D1, q3 weeks, Pre-Op & Post-Op (total 4 cycles)
  Interventions: Drug: Pre-operative chemotherapy
- Pre-operative concurrent chemoradiation therapy (Active Comparator)
  Interventions: Other: Pre-operative concurrent chemoradiation therapy

INTERVENTIONS:
Drug: Pre-operative chemotherapy — Docetaxel 75 mg/m2 + Carboplatin AUC(area under the curve)=6 on D1, q3 weeks, Pre-Op & Post-Op (total 4 cycles)
  Arms: Pre-operative chemotherapy
Other: Pre-operative concurrent chemoradiation therapy — Chemotherapy: Docetaxel 20 mg/m2 + carboplatin area under the curve = 2 on D1 and 8, q3weeks, Pre-Op & Post-Op: 2 cycles (total 4 cycles).
  Concurrent thoracic radiotherapy: Preoperative Thoracic radiation: 180cGy/fx, total: 4500cGy, 25fx
  Arms: Pre-operative concurrent chemoradiation therapy

SUMMARY:
This phase II trial is to compare neoadjuvant chemotherapy with concurrent chemoradiotherapy in patients with locally advanced non-small cell lung cancer (NSCLC) to address optimal induction strategy.

DETAILED DESCRIPTION:
Management of locally advanced non-small cell lung cancer (NSCLC) remains a challenge. Both local relapses and distant metastases are frequent, with 5-year survival of 3-17% for inoperable disease. Staging has historically subdivided stage III disease into clinical stage IIIA, thought to be potentially amenable to surgery, and stage IIIB, treated by defi nitive radiotherapy or radiochemotherapy. This phase II trial is to compare neoadjuvant chemotherapy with concurrent chemoradiotherapy in patients with locally advanced NSCLC to address optimal induction strategy.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologic diagnosis of non small-cell lung cancer
* Clinical stage IIIA and/or IIIB without pleural effusion
* ECOG functional status 0 or 1
* No renal function alteration (GFR >50%)
* No hepatic function alteration (ALT and AST less than 2 times its normal value)
* Leucocytes more than 2,000/mcl
* Hemoglobin more than 10mg/dL
* Platelets more than 100,000/mcl

Exclusion Criteria:

* Active uncontrolled infection.
* Serious concomitant disorders that would compromise the safety of patient or compromise the patient's ability to tolerate therapy.
* MI within preceding 6 months or symptomatic heart disease including unstable angina, congestive heart failure, or uncontrolled arrhythmia.
* Significant neurological or mental disorder.
* Second primary malignancy.
* Pregnant or nursing.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2007-02; Primary Completion 2011-01 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
To estimate the time to recurrence | Every 3 months

SECONDARY OUTCOMES:
To assess the pathologic complete response rate and the complete resection rate | Every 4 weeks
To estimate toxicities | Every 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jianxing He, MD, FACS, Principal Investigator — The First Affiliated Hospital of Guangzhou Medical University
Locations (1):
- The First Affiliated Hospital of Guangzhou Medical College, Guangzhou, Guangdong, China